CLINICAL TRIAL: NCT06159114
Title: Efficacy and Safety of Ningmitai Capsule Alone or Combined With Celecoxib in the Treatment of Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS): A Prospective, Randomized, Double-blind, Multicenter Clinical Study
Brief Title: Efficacy and Safety of Ningmitai Capsule Alone or Combined With Celecoxib in the Treatment of CP/CPPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xintian Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NM-23-A-006-YJ-006
Record Dates: First submitted 2023-11-19; First posted 2023-12-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Chronic Prostatitis
Keywords: NIH-CPSI; pain score; CP/CPPS
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ningmitai Capsule Group (Experimental): Patients take Ningmitai capsule, 0.38 g/capsule, tid, 4 capsules and celexcoib placebo, 0.2 g/ capsule, 1 capsule, qd each time, after meals, for 6 weeks.
  Interventions: Drug: Ningmitai capsule; Drug: Celecoxib placebo
- Celecoxib Capsule Group (Active Comparator): Patients take celexcoib capsule, 0.2 g/capsule, qd, 1 capsule and Ningmitai placebo, 0.38 g/ capsule, 4 cpsule, tid each time, after meals, for 6 weeks.
  Interventions: Drug: Celecoxib capsule; Drug: Ningmitai placebo
- Combined Group (Experimental): Patients take Ningmitai capsule, 0.38 g/capsule, tid, 4 capsules and celexcoib capsule, 0.2 g/ capsule, 1 capsule, qd each time, after meals, for 6 weeks.
  Interventions: Drug: Ningmitai capsule; Drug: Celecoxib capsule

INTERVENTIONS:
Drug: Ningmitai capsule — Ningmitai capsule (Ningmitai®) is Traditional Chinese Medicine which has already used in treatment of urinary system disease (eg. CPPS, BPH) in China for more than twenty years. The instruction of Ningmitai Capsule is 0.38g/capsule, 4 capsule/time, tid.
  Arms: Combined Group; Ningmitai Capsule Group
Drug: Celecoxib capsule — Celecoxib is one of NSAIDs recommended by the CUA Prostatitis Guidelines for alleviating pain symptoms in CP/CPPS patients. The instruction of Celecoxib capsule is 1 capsule at a time, 1 time a day.
  Arms: Celecoxib Capsule Group; Combined Group
Drug: Ningmitai placebo — Ningmitai placebo, a look-alike substance that contains no active drug, similar to Ningmitai capsule in color, smell, taste, shape, texture and other characteristics, 0.38g/ capsule.
  Arms: Celecoxib Capsule Group
Drug: Celecoxib placebo — Celecoxib placebo, a look-alike substance that contains no active drug, similar to Celecoxib capsule in color, smell, taste, shape, texture and other characteristics, 0.2g/ capsule.
  Arms: Ningmitai Capsule Group

SUMMARY:
1. Clinical trial title：Efficacy and safety of Ningmitai capsule alone or combined with celecoxib in the treatment of Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS): A prospective, randomized, double-blind, multicenter clinical study
2. Version number/date：1.1/2023-10-09
3. Principal investigator：Zhou Huiliang
4. Main research units：The First Affiliated Hospital of Fujian Medical University
5. Clinical trial start and end dates：2023/07/01-2025/12/31
6. Objective: To evaluate whether Ningmitai capsule(NMT) alone or combined with Celecoxib for 6 weeks is more effective than Celecoxib in improving pain symptoms of CP/CPPS patients.
7. Study type: Interventional study
8. Total sample size:240
9. Inclusion criteria:

（1）Age: male patients aged 18-60 years; （2）Long-term and repeated pelvic discomfort or pain (NIH-CPSI pain score ≥ 4 points), lasting more than 3 months, may be accompanied by different degrees of urination symptoms and sexual dysfunction; （3）Negative bacterial in urine before and after prostate massage; （4）Voluntarily participate in the trial. 10、Exclusion criteria:

1. Utilize any drugs for the treatment of chronic prostatitis in the past 2 weeks;
2. Patients who have received prostate surgery and treatment;
3. Urine WBC ≥ 5/HP, urinary system infection within 12 months, and effective antibiotic treatment in the early stage;
4. Pelvic pain and voiding dysfunction caused by non-prostatitis factors.
5. Suffering from serious primary cardiovascular disease, liver disease, kidney disease, hematological disease, lung disease or other serious diseases such as tumors or AIDS;
6. Significant adverse events in clinical or laboratory examination.
7. Allergic to the components of the test drugs or sulfa;
8. Previous active peptic ulcer / bleeding;
9. A birth plan within the past 8 months;
10. Legally disabled patients or psychiatric patients;
11. Suspected or confirmed alcohol or drug abuse, or other conditions that reduce the possibility of enrollment；
12. Participating in other clinical trials;
13. Considered unsuitable for enrollment by the investigator. 11、Interventions:

（1）Ningmitai group （2）Celecoxib group （3）Combination group

DETAILED DESCRIPTION:
1. Clinical trial title：Efficacy and safety of Ningmitai capsule alone or combined with celecoxib in the treatment of Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS): A prospective, randomized, double-blind, multicenter clinical study
2. Version number/date：1.1 /2023-10-09
3. Principal investigator：Zhou Huiliang
4. Main research units：The First Affiliated Hospital of Fujian Medical University
5. Clinical trial start and end dates：2023/07/01-2025/12/31
6. Objective: To evaluate whether using Ningmitai capsule(NMT) alone or combined with Celecoxib for 6 weeks is more effective than Celecoxib in improving symptoms especially pain of CP/CPPS patients.
7. Study type: Interventional study
8. Total sample size: 240
9. Inclusion criteria:

(1)Age: male patients aged 18-60 years; (2)Long-term and repeated pelvic discomfort or pain (NIH-CPSI pain score ≥ 4 points), lasting more than 3 months, may be accompanied by different degrees of urination symptoms and sexual dysfunction; (3)Negative bacterial in urine before and after prostate massage; (4)Voluntarily participate in the trial and agree to sign an informed consent form.

10、Exclusion criteria:

(1)Use any non-steroidal anti-inflammatory drugs，α receptor blockers，antibiotics, PDE5 inhibitors or other traditional Chinese medicines or botanicals for the treatment of prostatitis in the past 2 weeks; those who are using drugs for the treatment of prostatitis need to stop the drug for 2 weeks before the clinical trial; (2)Patients who have received prostate surgery and treatment such as TURP, TUIP, open prostatectomy, biofeedback therapy, hyperthermia, ablation, prostate cryotherapy, transperineal extracorporeal shock wave therapy, prostate injection therapy, transurethral prostate perfusion therapy, or bladder surgery such as bladder neck incision; (3)Urine WBC ≥ 5 /HP, urinary system infection within 3 months; (4)Pelvic pain and voiding dysfunction caused by non-prostatitis factors, such as benign prostatic hyperplasia, diseases of testis, epididymis and spermatic cord, overactive bladder, neurogenic bladder, interstitial cystitis, glandular cystitis, sexually transmitted diseases, bladder tumor, prostate cancer, anorectal disease, lumbar disease, central and peripheral neuropathy; (5)Suffering from serious primary cardiovascular disease, liver disease, kidney disease, hematological disease, lung disease or other serious diseases such as tumors or AIDS; (6)Significant adverse events in clinical or laboratory examination indicators, such as ALT and AST ≥ 1.5 times the upper limit of reference value, creatinine (SCR) > the upper limit of reference value; (7)Allergic to the components of the test drugs or sulfa; (8)Previous active peptic ulcer / bleeding; (9)A birth plan within the past 8 months; (10)Legally disabled patients (blind, deaf, mute, intellectual disability, etc.), psychiatric patients; (11)Suspected or confirmed alcohol or drug abuse, or other conditions that reduce the possibility of enrollment or complicate enrollment according to the judgment of the investigator, such as frequent changes in the working environment that are likely to cause loss to follow-up; (12)Participating in other clinical trials; (13)Considered unsuitable for enrollment by the investigator. 11、Interventions:

1. Ningmitai group Orally administered Ningmitai capsule and Celecoxib placebo after meals for 6 weeks.

   Ningmitai capsule: 0.38 g/capsule, tid, 4 capsules each time; Celecoxib placebo: 0.2 g/capsule, qd，1 capsule each time. Sample size: 80
2. Celecoxib group Orally administered Celecoxib capsule and Ningmitai placebo after meals for 6 weeks.

   Celecoxib capsule: 0.2 g/capsule, qd，1 capsule each time; Ningmitai placebo: 0.38 g/capsule, tid, 4 capsules each time. Sample size: 80
3. Combination group Orally administered Ningmitai capsule and Celecoxib capsule after meals for 6 weeks.

Ningmitai capsule: 0.38 g/capsule, tid, 4 capsules each time; Celecoxib capsule: 0.2 g/capsule, qd，1 capsule each time. Sample size: 80 12、Treatment cycle：6 weeks. the trial treatment began on the day of randomization.

13、Visiting nodes：① before treatment (-2 weeks to 0 days), ②2 weeks of treatment (14 ± 2 days), ③ 4 weeks of treatment (28 ± 5 days).④ 6 weeks of treatment（42 ± 7 days).

14、Countries of recruitment and research settings: Country:China Province:Fujian Institutions (hospitals): The First Affiliated Hospital of Fujian Medical University, The First Affiliated Hospital of Xiamen University.

15、Recruiting status: Not yet recruiting 16、Randomization Procedure:In this study, the research center was used as the stratification factor of random assignment. Subjects were randomly assigned (1:1:1) to NMT group, Celecoxib group and combination group according to the random allocation table (subject random code) simulated by SAS 9.2 software. Subjects' random numbers cannot be reused by other subjects, whether they are using the study drug or not, or the study is terminated for any reason.

17、Sign the informed consent: Yes. 18、Data collection and Management (A standard data collection and management system include a CRF and an electronic data capture:In this study, case report form (CRF) was used to collect and manage research data. The sponsor or designated person is responsible for data management of the study, including data quality control. The workflow of data management includes data entry, data verification and query, medical coding, data audit, database locking, data export and transmission, data and data management file archiving, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age: male patients aged 18-60 years;
2. Long-term and repeated pelvic discomfort or pain (NIH-CPSI pain score ≥ 4 points), lasting more than 3 months, may be accompanied by different degrees of urination symptoms and sexual dysfunction;
3. Negative bacterial in urine before and after prostate massage;
4. Voluntarily participate in the trial and agree to sign an informed consent form.

Exclusion Criteria:

1. Use any non-steroidal anti-inflammatory drugs，α receptor blockers，antibiotics, PDE5 inhibitors or other traditional Chinese medicines or botanicals for the treatment of prostatitis in the past 2 weeks; those who are using drugs for the treatment of prostatitis need to stop the drug for 2 weeks before the clinical trial;
2. Patients who have received prostate surgery and treatment such as TURP, TUIP, open prostatectomy, biofeedback therapy, hyperthermia, ablation, prostate cryotherapy, transperineal extracorporeal shock wave therapy, prostate injection therapy, transurethral prostate perfusion therapy, or bladder surgery such as bladder neck incision;
3. Urine WBC ≥ 5 /HP, urinary system infection within 3 months;
4. Pelvic pain and voiding dysfunction caused by non-prostatitis factors, such as benign prostatic hyperplasia, diseases of testis, epididymis and spermatic cord, overactive bladder, neurogenic bladder, interstitial cystitis, glandular cystitis, sexually transmitted diseases, bladder tumor, prostate cancer, anorectal disease, lumbar disease, central and peripheral neuropathy;
5. Suffering from serious primary cardiovascular disease, liver disease, kidney disease, hematological disease, lung disease or other serious diseases such as tumors or AIDS;
6. Significant adverse events in clinical or laboratory examination indicators, such as ALT and AST ≥ 1.5 times the upper limit of reference value, creatinine (SCR) > the upper limit of reference value;
7. Allergic to the components of the test drugs or sulfa;
8. Previous active peptic ulcer / bleeding;
9. A birth plan within the past 8 months;
10. Legally disabled patients (blind, deaf, mute, intellectual disability, etc.), psychiatric patients;
11. Suspected or confirmed alcohol or drug abuse, or other conditions that reduce the possibility of enrollment or complicate enrollment according to the judgment of the investigator, such as frequent changes in the working environment that are likely to cause loss to follow-up;
12. Participating in other clinical trials;
13. Considered unsuitable for enrollment by the investigator.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 246 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Pain score of the National Institutes of Health Chronic Prostatitis Symptom Index | Treatment for 6 weeks
  The change of NIH-CPSI pain score from baseline to 6 weeks. National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.

SECONDARY OUTCOMES:
Pain score of the National Institutes of Health Chronic Prostatitis Symptom Index | Treatment for 2 weeks
  The change of NIH-CPSI pain score from baseline to 2 weeks，respectively. National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.
Pain score of the National Institutes of Health Chronic Prostatitis Symptom Index | Treatment for 4 weeks
  The change of NIH-CPSI pain score from baseline to 4 weeks，respectively. National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.
Total score, urinary score and quality of life score of the National Institutes of Health Chronic Prostatitis Symptom Index | Treatment for 2 weeks
  The change of NIH-CPSI total score, urinary score and quality of life score from baseline to 2 weeks. National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.
Total score, urinary score and quality of life score of the National Institutes of Health Chronic Prostatitis Symptom Index | Treatment for 4 weeks
  The change of NIH-CPSI total score, urinary score and quality of life score from baseline to 4 weeks. National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.
Total score, urinary score and quality of life score of the National Institutes of Health Chronic Prostatitis Symptom Index | Treatment for 6 weeks
  The change of NIH-CPSI total score, urinary score and quality of life score from baseline to 6 weeks. National Institutions of Health Chronic Prostatitis Symptom Index（NIH-CPSI，0~43 points） consists of three subscales. The first part is pain symptoms, which consists of questions 1~4 (0~21 points), and evaluates the location, frequency and severity of pain. The second part is urination symptoms, which consists of questions 5~6 (0 ~ 10 points), and evaluates the severity of incomplete urination and frequent urination; The third part is to evaluate the impact on the quality of life, which consists of questions 7~9 (0~12 points).The higher the score, the more serious the symptoms of chronic prostatitis.
The scores of questions 1~4 of the National Institutes of Health Chronic Prostatitis Symptom Index | Treatment for 2 weeks
  The change of scores of NIH-CPSI questions 1~4 from baseline to 2 weeks. Questions 1~4 (0~21 points) evaluates the location, frequency and severity of pain. The higher the score, the more serious the pain symptoms of chronic prostatitis.
The scores of questions 1~4 of the National Institutes of Health Chronic Prostatitis Symptom Index | Treatment for 4 weeks
  The change of scores of NIH-CPSI questions 1~4 from baseline to 4 weeks. Questions 1~4 (0~21 points) evaluates the location, frequency and severity of pain. The higher the score, the more serious the pain symptoms of chronic prostatitis.
The scores of questions 1~4 in the National Institutes of Health Chronic Prostatitis Symptom Index | Treatment for 6 weeks
  The change of scores of questions 1~4 in NIH-CPSI from baseline to 6 weeks. Questions 1~4 (0~21 points) evaluates the location, frequency and severity of pain. The higher the score, the more serious the pain symptoms of chronic prostatitis.
Response rate | Treatment for 2 weeks, 4 weeks and 8 weeks
  The response rate is defined as a decrease of at least 2 points in the NIH-CPSI pain score and at least 4 points in the NIH-CPSI total score, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No